CLINICAL TRIAL: NCT04776057
Title: Rotation Stability of Toric Intraocularlens (IOL) Compared Sitting Against Lying After Cataract Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof Oliver Findl, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 20-302-1220
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lying (Other): after cataract lying for 1 hour
  Interventions: Other: catarct surgery with toric intra ocular lenses
- sitting, walkin (Other): after cataract sitting or walking for 1 hour
  Interventions: Other: catarct surgery with toric intra ocular lenses

INTERVENTIONS:
Other: catarct surgery with toric intra ocular lenses — rotation stability of toric intraocular lenses between sitting or routine settings (sitting, going around) after cataract operation

SUMMARY:
To assess the rotation stability of toric intraocular lenses between sitting or routine settings (sitting, going around) after cataract operation.

DETAILED DESCRIPTION:
To assess the rotation stability of toric intraocular lenses between sitting or routine settings (sitting, going around) after cataract operation.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Regular corneal astigmatism ≥ 1.5 D
* written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as: pseudoexfoliation, traumatic cataract corneal scars, and other co-morbidity that could affect capsule bag stability ( e.g. Marfan syndrome)
* High myopia (> 29 mm AL)
* Irregular corneal astigmatism on corneal topography
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of toric IOL rotation between both groups (mean ≠ SD) | 1 Year
  Aim is to see if the lying down after the operation lowers the risk of toric IOL rotation compared to sitting down

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria